CLINICAL TRIAL: NCT01028183
Title: Impact of Maternal-infant Therapeutics on Safety, Mortality, and Disability
Status: Withdrawn | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Daniel K Benjamin Jr MD PhD MPH, Associate Professor of Pediatrics, Duke Clinical Research Institute
Other Study IDs: IRB pending
Record Dates: First submitted 2009-12-05; First posted 2009-12-09 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Gastroesophageal Reflux; Presumed Sepsis; Patent Ductus Arteriosus; Chronic Lung Disease; Neurodevelopmental Impairment
Keywords: therapeutics; safety; maternal; neonatal
MeSH Terms: conditions — Gastroesophageal Reflux; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Extremely Premature Infants: < 30 weeks gestation (N=5000)
- Premature Infants: 30-36 weeks gestation (N=2000)
- Hospitalized Term Infants: >=37 weeks gestation (N=2000)
- Healthy Term Infants: >=37 weeks gestation (N=1000)

SUMMARY:
The purpose of this research is to address the comparative effectiveness and harm of the therapeutics frequently given to pregnant women and their young infants including antibiotics, tocolytic agents, non-steroidal anti-inflammatory drugs, H2 blockers, and steroids.

Our overall hypothesis is that the use of an existing electronic medical record with additional resources for precise data collection and 18 month follow up will successfully address current knowledge gaps in therapeutic effectiveness and relative therapeutic harm.

We will use an existing electronic medical record into which detailed healthcare information is entered for over 100,000 newborns each year. These infants will comprise the "Source Cohort". Nested within that database, we will prospectively enroll 10% of the population (10,000 newborns) as the Follow-Up Cohort.

The current electronic medical record for the Source Cohort does not capture therapeutic dosing with sufficient precision to conduct comparative effectiveness research sufficient to change medical practice. The proposed research will: 1) ensure accurate data collection through electronic monitoring and real-time quality assurance evaluation in the Source Cohort; and 2) conduct 18 months post-hospital follow-up for neurologic outcomes and disability for the Follow-Up Cohort. We will complete assessments of neurologic outcomes and disability using an interactive web-based system, mail, telephone follow up, and in-person examination.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the a Pediatrix Medical Group NICU
* <=5 days of life
* likely to follow-up at 18 months adjusted age

Exclusion Criteria:

* failure to consent

Max Age: 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will enroll 10,000 infants at 40 centers. Infants will be enrolled into one of four strata: extremely premature (<30 weeks, n=5,000), premature (30-36 weeks inclusive n=2,000), hospitalized term (≥37 weeks gestation, n=2,000), and healthy term (≥37 weeks gestation, n=1,000).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Estimated); Study Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Benjamin, MD PhD MPH, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States